CLINICAL TRIAL: NCT03725761
Title: A Multi-arm, Phase 2 Study to Evaluate the Safety and Efficacy of Sacituzumab Govitecan in Patients With Metastatic Castration-Resistant Prostate Cancer Who Have Progressed on Second Generation AR-Directed Therapy
Brief Title: Sacituzumab Govitecan in Patients With Metastatic Castration-Resistant Prostate Cancer Progressing on Second Generation AR-Directed Therapy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW18043; P30CA014520 (NIH); A534260 (Other: UW Madison); SMPH\MEDICINE\HEM-ONC (Other: UW Madison); NCI-2018-02551 (Registry Identifier: NCI Trial ID); Protocol Version 5/12/2022 (Other: UW Madison); 2018-0857 (Other: UW-Madison IRB)
Record Dates: First submitted 2018-10-15; First posted 2018-10-31 (Actual); Results first posted 2025-04-24 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Prostate Cancer
Keywords: Prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — sacituzumab govitecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sacituzumab Govitecan Treatment (Experimental): Subjects enrolled in this study will receive Sacituzumab Govitecan in addition to their single agent Androgen Receptor Signaling Inhibitors (ARSI) as treatment for Castrate-Resistant Prostate Cancer. Dose will be calculated per protocol in milligrams based on the subject's body weight at the beginning of each cycle or more frequently if weight changes >10%. Subjects will be treated on days 1 and 8 in a 21-day cycle, minimum 3 cycles.
  Interventions: Drug: Sacituzumab Govitecan

INTERVENTIONS:
Drug: Sacituzumab Govitecan — Sacituzumab Govitecan is a novel Antibody Drug Conjugate (ADC) based on a humanized anti-Trop-2 antibody (hRS7) conjugated to SN-38 payload.
  Other Names: IMMU-132

SUMMARY:
This study will investigate the safety and efficacy of Sacituzumab Govitecan in patients with metastatic castration-resistant prostate cancer progressing on second generation androgen receptor (AR) directed therapy (e.g., enzalutamide, darolutamide, apalutamide and/or abiraterone).

DETAILED DESCRIPTION:
This study will investigate the safety and efficacy of Sacituzumab Govitecan in patients with metastatic castration-resistant prostate cancer progressing on second generation AR-directed therapy. Patients who have progressed while on therapy with combination enzalutamide/abiraterone or ARN-509/abiraterone as part of ongoing clinical trials are allowed and may be enrolled in the study. To better understand the heterogeneity of response and in particular to identify patients likely to benefit, an extensive correlative biomarker program will be included to collect and analyze tumor tissue biopsies, circulating tumor cells (CTCs), and circulating tumor DNA (ctDNA).

A validated predictive biomarker would benefit the individual patient by enabling him to be treated with a safe effective oral drug and avoid one from which he is unlikely to benefit. It is also essential for prostate cancer drug development because the increasing availability of more life-prolonging therapies is making it more difficult to prove a survival benefit for the next promising agent.

ELIGIBILITY:
Inclusion Criteria:

* Documented histological or cytological evidence of adenocarcinoma of the prostate
* Documented metastatic disease on bone scan and/or CT scans
* Currently receiving enzalutamide, darolutamide, apalutamide and/or abiraterone. Subjects who have received combination enzalutamide/abiraterone or combination apalutamide/abiraterone as part of clinical trials are allowed but will need to be receiving only a single agent ARSI at the time of study enrollment. Subjects who have received any other therapeutic investigational product directed towards the AR or androgen biosynthesis are allowed. Prior treatment with first-generation AR antagonists (i.e., bicalutamide, nilutamide, flutamide) before second generation AR-directed therapy is allowed.
* Demonstrated disease progression while on enzalutamide, darolutamide, apalutamide, and/or abiraterone. Progressive disease is defined by one or more of the following:

  * A rise in prostate specific antigen (PSA) on two successive determinations at least one week apart and PSA level ≥2 ng/mL
  * Soft-tissue progression defined by RECIST 1.1
  * Bone disease progression defined by Prostate Cancer Working Group 2 (PCWG2) with ≥2 new lesions on bone scan
* A minimum serum PSA level of ≥2 ng/mL that is rising based on the PCWG2 criteria
* ≥18 y ears of age
* Castrate levels of testosterone (<50 ng/dL [1.74 nmol/L])
* Undergone orchiectomy, or have been on Luteinizing hormone-releasing hormone (LHRH) agonists or antagonists, for at least 3 months prior to study treatment start. Subjects on LHRH agonists/antagonists must remain on these agents for the duration of the study
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1
* Normal organ function with acceptable initial laboratory values within 30 days of study treatment start:

  * White Blood Cell Count (WBC) greater than or equal to 3000/μl
  * Absolute Neutrophil Count (ANC) greater than or equal to 1000/μl
  * Platelet count greater than or equal to100,000/μl
  * Hemoglobin (HGB) greater than or equal to 9 g/dL
* Adequate hepatic function as evidenced by Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels less than 3X the upper limit of normal (ULN) and bilirubin levels of less than 2.0 mg/dl.
* Adequate renal function as evidenced by serum creatinine of less than 2.0 mg/dL
* Able to provide written informed consent, or have a legal representative provide written informed consent
* Subjects must have a previously-acquired biopsy from a metastatic site available
* Subjects must be willing and able (in the opinion of the treating physician) to undergo one research biopsy for the investigational component of this study
* Subjects who have partners of child-bearing potential must be willing to use at least two forms of effective birth control (one form must be a barrier method) during the treatment period and for 90 days after last dose of IMMU-132. Subjects must also agree to not donate sperm through 90 days following the last dose of IMMU-132.

Exclusion Criteria:

* Received prior cytotoxic chemotherapy such as docetaxel, cabazitaxel or platinum chemotherapy for metastatic prostate cancer, castration sensitive or castration resistant, within two years prior to study entry. Neoadjuvant chemotherapy is allowed.
* Completed sipuleucel-T (Provenge ®) treatment within 30 days of study treatment start.
* Received any therapeutic investigational agent within 2 weeks of study treatment start.
* Received palliative radiotherapy within 4 weeks of study treatment start.
* Received herbal products or alternative therapies that may decrease PSA levels or that may have hormonal anti-prostate cancer activity (e.g., saw palmetto, PC-SPES, PC-HOPE, St. John's wort, selenium supplements, grape seed extract, etc.) within 4 weeks of study treatment start or plans to initiate treatment with these products/alternative therapies during the entire duration of the study.
* Active central nervous system (CNS) metastases from prostate cancer. Subjects with treated epidural disease are eligible to enroll. Subjects with treated brain metastases can be included as long as >4 weeks have elapsed since last treatment (radiotherapy or surgery) for brain metastases, the subject is neurologically and radiographically stable, and is not receiving corticosteroids for brain metastases. Subjects with untreated brain metastases are excluded. Brain imaging (CT or MRI) is not required at baseline if brain metastases are not clinically suspected.
* A history within the last 3 years of another invasive malignancy (excluding non-melanoma skin cancer).
* A QTcF interval of >470 msec on the initial Screening ECG; if the Screening ECG QTcF interval is >470 msec, then it may be repeated two more times, and if the mean QTcF of the 3 ECGs is ≤470 msec, the subject may be enrolled.
* A history of clinically significant cardiac arrhythmias including ventricular tachycardia, ventricular fibrillation, torsades de pointes and second degree or third degree atrioventricular heart block without a permanent pacemaker in place. Subjects with resolved or rate-controlled atrial fibrillation/atrial flutter are allowed.
* NYHA Class III or IV congestive heart failure, unstable angina, myocardial infarction/acute coronary syndrome within the preceding 6 months.
* Diabetes mellitus with more than 2 episodes of diabetic ketoacidosis in the 12 months preceding study treatment start.
* Inadequately controlled hypertension (defined as blood pressure >150mmHg systolic and/or >100 mmHg diastolic despite antihypertensive medication) or any history of hypertensive crisis or hypertensive encephalopathy.
* History of loss of consciousness or transient ischemic attack within 12 months before study treatment start.
* Known active HIV, Hepatitis B, or Hepatitis C infections.
* Any other medical, psychiatric, or social condition, including substance abuse, which in the opinion of the Investigator would preclude safe participation in the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-10-24 (Actual); Primary Completion 2024-04-18 (Actual); Study Completion 2027-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Lang, MD, Principal Investigator — University of Wisconsin, Madison
Locations (3):
- United States (3):
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Weill Cornell Medical College, New York, New York
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/

RESULTS

PARTICIPANT FLOW:
Groups:
- Sacituzumab Govitecan Treatment: Participants enrolled in this study will receive Sacituzumab Govitecan in addition to their single agent Androgen Receptor Signaling Inhibitors (ARSI) as treatment for Castrate-Resistant Prostate Cancer. Dose will be calculated per protocol in milligrams based on the participant's body weight at the beginning of each cycle or more frequently if weight changes >10%. Participants will be treated on days 1 and 8 in a 21-day cycle, minimum 3 cycles.
  Sacituzumab Govitecan is a novel Antibody Drug Conjugate (ADC) based on a humanized anti-Trop-2 antibody (hRS7) conjugated to SN-38 payload.
Period: Overall Study
Arm/Group | Sacituzumab Govitecan Treatment
Started | 31
Received Treatment | 31
Off Study Treatment Early | 11
Completed Treatment (At least 9 weeks study treatment is defined as completed treatment) | 19
Currently on Treatment | 1
Completed (participants followed until progression, initiation of new anti-cancer therapy, or death) | 30
Not Completed | 1
Not completed — still on study | 1

BASELINE CHARACTERISTICS:
Groups:
- Sacituzumab Govitecan Treatment: Participants enrolled in this study will receive Sacituzumab Govitecan in addition to their single agent ARSI as treatment for Castrate-Resistant Prostate Cancer. Dose will be calculated per protocol in milligrams based on the participant's body weight at the beginning of each cycle or more frequently if weight changes >10%. Participants will be treated on days 1 and 8 in a 21-day cycle, minimum 3 cycles.
Arm/Group | Sacituzumab Govitecan Treatment
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (8.0)
Age, Customized [Count of Participants; unit: Participants]
  50-59 years | 5
  60-69 years | 12
  70-79 years | 10
  80-89 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 25
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 31
Baseline Prostate Specific Antigen (PSA) [Median (Full Range); unit: ng/ml] | 30 [3 to 3852]
History of Chemotherapy [Count of Participants; unit: Participants]
  Chemo Naive | 25
  Chemo Exposed | 6

OUTCOME MEASURES:

1. Primary Outcome: PSA Response Rate
Description: Subjects who achieve ≥50% PSA decline at or before 9 weeks of therapy with Sacituzumab Govitecan (IMMU-132) are considered to have responded. PSA responses will be analyzed by descriptive statistics and summarized in tabular format (frequency tables). The overall PSA response rate will be reported along with the corresponding 95% confidence interval which will be constructed using the Wilson score method.
Time Frame: up to 9 weeks
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Sacituzumab Govitecan Treatment
Number analyzed (Participants) | 31
percent | 6 [2 to 21]

2. Primary Outcome: 6-Month Progression Free Survival Rate
Description: Proportion of participants remaining alive and progression free (using Prostate Cancer Working Group 2 (PCWG2) criteria) 6 months from time of starting treatment as estimated by the Kaplan-Meier method.
Time Frame: 6 months
Measure: Number; unit: percent
Arm/Group | Sacituzumab Govitecan Treatment
Number analyzed (Participants) | 31
percent | 52

3. Secondary Outcome: Median Progression Free Survival Rate
Description: The probability distribution of Progression Free Survival (PFS) will be estimated using the Kaplan-Meier method. The median will be estimated from this distribution. Subjects who have not died or progressed (using PCWG2 criteria) will be censored at the date of last assessment.
Time Frame: Up to 2 years from start of treatment
Reporting Status: Not Posted

4. Secondary Outcome: Radiologic Response Rate
Description: The number of participants with progressive disease, stable disease, partial response and complete response will be summarized in tabular format. The overall response rate will be reported along with the corresponding 95% confidence interval which will be constructed using the Wilson score method.
Time Frame: up to 2 years from start of treatment
Reporting Status: Not Posted

5. Secondary Outcome: Median Overall Survival
Description: Overall Survival (OS) is the duration from start of treatment until death from any cause. The probability distribution of OS will be estimated using the Kaplan-Meier method. The median will be estimated from this distribution. Subjects who have not died will be censored at the date of last contact.
Time Frame: Up to 2 years from start of treatment
Reporting Status: Not Posted

6. Secondary Outcome: Toxicity Rates (Grade 2, Grade 3, Grade 4, Grade ≥ 2, Grade ≥ 3, Etc.)
Description: Toxicities will be summarized by type and severity in tabular format. Toxicity rates (Grade 2, Grade 3, Grade 4, Grade ≥ 2, Grade ≥ 3, etc.) will be calculated and reported along the corresponding 95% confidence intervals. The 95% confidence intervals will be constructed using the Wilson score method.
Time Frame: Up to 9 weeks from start of treatment
Measure: Count of Units; unit: number of adverse events
Units Other Than Participants: number of adverse events
Groups:
- Grade 2; Greater Than or Equal to 2: Grade 2 is a moderate level of toxicity per the Common Toxicity Criteria scale from Grade 0 (no toxicity) to Grade 5 (death).
- Grade 3; Greater Than or Equal to 3: Grade 3 is a severe level of toxicity per the Common Toxicity Criteria scale from Grade 0 (no toxicity) to Grade 5 (death).
- Grade 4; Greater Than or Equal to 4: Grade 4 is a life-threatening level of toxicity per the Common Toxicity Criteria scale from Grade 0 (no toxicity) to Grade 5 (death).
Arm/Group | Grade 2 | Grade 3 | Grade 4 | Greater Than or Equal to 2 | Greater Than or Equal to 3 | Greater Than or Equal to 4
Number analyzed (Participants) | 31 | 31 | 31 | 31 | 31 | 31
Number analyzed (number of adverse events) | 73 | 31 | 11 | 115 | 42 | 11
number of adverse events
  Alopecia | 10 | 0 | 0 | 10 | 0 | 0
  Anemia | 8 | 4 | 0 | 12 | 4 | 0
  Anorexia | 4 | 0 | 0 | 4 | 0 | 0
  Creatinine increased | 1 | 0 | 0 | 1 | 0 | 0
  Dehydration | 1 | 0 | 0 | 1 | 0 | 0
  Diarrhea | 8 | 7 | 0 | 15 | 7 | 0
  Dysgeusia | 1 | 0 | 0 | 1 | 0 | 0
  Dyspnea | 1 | 0 | 0 | 1 | 0 | 0
  Fatigue | 5 | 0 | 0 | 5 | 0 | 0
  Febrile neutropenia | 0 | 2 | 0 | 2 | 2 | 0
  Hyponatremia | 1 | 0 | 0 | 1 | 0 | 0
  Hypophosphatemia | 1 | 0 | 0 | 1 | 0 | 0
  Infusion site extravasation | 1 | 0 | 0 | 1 | 0 | 0
  Intermittent body aches, general | 1 | 0 | 0 | 1 | 0 | 0
  Mucositis oral | 1 | 0 | 0 | 1 | 0 | 0
  Muscle weakness lower limb | 1 | 0 | 0 | 1 | 0 | 0
  Nausea | 5 | 1 | 0 | 6 | 1 | 0
  Neutrophil count decreased | 9 | 12 | 7 | 28 | 19 | 7
  Peripheral ischemia | 1 | 0 | 0 | 1 | 0 | 0
  Platelet count decreased | 1 | 0 | 0 | 1 | 0 | 0
  Rash maculo-papular | 4 | 0 | 0 | 4 | 0 | 0
  Sinus tachycardia | 1 | 0 | 0 | 1 | 0 | 0
  Syncope | 0 | 1 | 0 | 1 | 1 | 0
  Typhlitis | 0 | 1 | 0 | 1 | 1 | 0
  Vasovagal reaction | 0 | 1 | 0 | 1 | 1 | 0
  White blood cell decreased | 7 | 2 | 4 | 13 | 6 | 4

ADVERSE EVENTS:
Time Frame: up to 6 months
Arm/Group | Sacituzumab Govitecan Treatment
All-Cause Mortality (participants affected / at risk) | 30/31
Serious Adverse Events (participants affected / at risk) | 12/31
Other Adverse Events (participants affected / at risk) | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sacituzumab Govitecan Treatment (N=31)
Spinal Cord Compression (Nervous system disorders) | 3
Bladder Infection (Infections and infestations) | 1
Typhlitis (Gastrointestinal disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 2
Syncope (Nervous system disorders) | 1
Atrial Flutter (Cardiac disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Myocardial infarction (Cardiac disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sacituzumab Govitecan Treatment (N=31)
Anemia (Blood and lymphatic system disorders) | 17 (31)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1)
Heart Failure (Cardiac disorders) | 1 (1)
Sinus Tachycardia (Cardiac disorders) | 1 (1)
Adrenal Insufficiency (Endocrine disorders) | 1 (1)
Chills (General disorders) | 3 (3)
Debility (General disorders) | 1 (1)
Edema Limbs (General disorders) | 2 (2)
Fatigue (General disorders) | 13 (17)
Fever (General disorders) | 1 (1)
Gait Disturbance (General disorders) | 3 (3)
Generalized Weakness (General disorders) | 2 (2)
Hernia (General disorders) | 1 (1)
Infusion Site Extravasation (General disorders) | 1 (1)
Injection Site Reaction (General disorders) | 1 (1)
Localized Edema (General disorders) | 2 (2)
Non-Cardiac Chest Pain (General disorders) | 2 (2)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) — Intermittent Body Aches
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) — Fluid collection in the presacral space
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) — Lassitude
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) — Worsening Chronic Pain
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 12 (17)
Diarrhea (Gastrointestinal disorders) | 20 (41)
Dry Mouth (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 2 (2)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Mucositis Oral (Gastrointestinal disorders) | 1 (3)
Nausea (Gastrointestinal disorders) | 19 (34)
Stomach Pain (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 9 (19)
Gastrointestinal disorders other, specify (Gastrointestinal disorders) | 1 (1) — belching
Gastrointestinal disorders other, specify (Gastrointestinal disorders) | 1 (1) — Loose Stools
Gastrointestinal disorders other, specify (Gastrointestinal disorders) | 1 (1) — Left Groin Hernia
Bronchial Infection (Infections and infestations) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1)
Lip Infection (Infections and infestations) | 1 (1)
Rash Pustular (Infections and infestations) | 1 (1)
Rhinitis Infective (Infections and infestations) | 2 (2)
Urinary Tract Infection (Infections and infestations) | 2 (2)
Upper Respiratory Infection (Infections and infestations) | 3 (3)
Infections and infestations - Other, specify (Infections and infestations) | 2 (2) — COVID-19
Fall (Injury, poisoning and procedural complications) | 3 (3)
Alanine aminotransferase increased (Investigations) | 2 (2)
Alkaline phosphatase increased (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 3 (3)
Blood bilirubin increased (Investigations) | 1 (1)
Cardiac troponin T increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 3 (5)
Neutrophil count decreased (Investigations) | 20 (38)
Platelet count decreased (Investigations) | 7 (12)
Weight Loss (Investigations) | 3 (3)
White blood cell decreased (Investigations) | 12 (23)
Investigations - Other,specify (Investigations) | 1 (1) — protein total decreased
Anorexia (Metabolism and nutrition disorders) | 14 (14)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 8 (13)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 11 (12)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 3 (4)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 7 (7)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 6 (11)
Bone Pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 5 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 3 (4)
Weakness in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorders -Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) — Knee pain
Musculoskeletal and connective tissue disorders -Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) — Left Hip Pain
Musculoskeletal and connective tissue disorders -Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) — Iliac Pain
Musculoskeletal and connective tissue disorders -Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) — Left hip and leg pain
Musculoskeletal and connective tissue disorders -Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) — Left Rib Pain
Musculoskeletal and connective tissue disorders -Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) — Discomfort in left clavicle
Dizziness (Nervous system disorders) | 5 (5)
Dysgeusia (Nervous system disorders) | 3 (3)
Headache (Nervous system disorders) | 3 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2)
Presyncope (Nervous system disorders) | 1 (1)
Spinal Cord Compression (Nervous system disorders) | 1 (1)
Vasovagal Reaction (Nervous system disorders) | 1 (1)
Memory Impairment (Nervous system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Epitaxis (Respiratory, thoracic and mediastinal disorders) | 2 (5)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Dry Nasal
Genital Edema (Reproductive system and breast disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (3)
Hematuria (Renal and urinary disorders) | 3 (3)
Incomplete continence (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Urinary Frequency (Renal and urinary disorders) | 1 (1)
Urinary Incontinence (Renal and urinary disorders) | 2 (2)
Urinary Tract Pain (Renal and urinary disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 18 (22)
Dry Skin (Skin and subcutaneous tissue disorders) | 3 (3)
Pruritis (Skin and subcutaneous tissue disorders) | 3 (3)
Rash - Delayed Hypersensitivity Reaction (rash on neck, flank, leg) (Skin and subcutaneous tissue disorders) | 1 (1)
Rash Maculo-papular (Skin and subcutaneous tissue disorders) | 6 (10)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) — Scalp Itchiness
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) — Small Lump on Scalp
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) — Left Forearm Lesion
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) — rash
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1 (1) — Port placement
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1 (1) — Right Femur TFNA
Hot Flashes (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 3 (4)
Hypotension (Vascular disorders) | 3 (3)
Thromborembolic event (Vascular disorders) | 1 (1)
Peripheral Ishcemia (Vascular disorders) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 1 (1) — Itchy Eyes

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-12): https://cdn.clinicaltrials.gov/large-docs/61/NCT03725761/Prot_SAP_000.pdf